CLINICAL TRIAL: NCT01365130
Title: A Phase II Study Of Cabazitaxel For Metastatic Gastroesophageal Adenocarcinomas That Have Relapsed After At Least One Line Of Chemotherapy
Brief Title: Chemotherapy for Patients With Gastroesophageal Cancers Who Have Progressed After One Prior Chemo Regimen
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: As of 12/12/12 study closed to enrollment because study was determined to be ineffective.
Sponsor: howard safran (Other)
Collaborators: Roger Williams Medical Center (Other); Rhode Island Hospital (Other); The Miriam Hospital (Other)
Responsible Party: Sponsor-Investigator, howard safran, Priniciple Investigator, Brown University
Organization: Brown University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 243
Record Dates: First submitted 2011-05-11; First posted 2011-06-03 (Estimated); Results first posted 2014-04-28 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Esophageal; Gastrooesophageal Cancer; Gastric Cancer
Keywords: esophageal cancer; gastroesophageal cancer; gastric cancer
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms | interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- real drug (Experimental): patients will receive Jevtana 25mg/m2, IV every 21 days until disease progression or unacceptable toxicity
  Interventions: Drug: jevtana

INTERVENTIONS:
Drug: jevtana — Cabazitaxel 25mg/m2, IV every 21 days until progression
  Other Names: Cabazitaxel

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Cabazitaxel, as well as safety and side effects for patients with advanced gastroesophageal cancer

DETAILED DESCRIPTION:
Gastric cancer is the second most frequent cancer-related cause of death after lung cancer worldwide with approximately 900,000 cases per year. The incidence of gastric cancer is highest in East Asia, China and Japan. In the last two decades there has been a dramatic increase in North America and Europe of adenocarcinoma of the distal esophagus and GE junction which are indistinguishable from proximal gastric cancer.

Cabazitaxel (XRP6258) is a semi-synthetic novel taxoid. Like traditional taxane drugs, it binds to and stabilizes tubilin structures resulting in inhibition of cold-induced microtubule depolymerization and cell division with subsequent inhibition of tumor cell proliferation. This novel agent, however, has poor affinity for P-glycoprotein--the protein product of multidrug resistance gene ABCB1. P-glycoprotein is a membrane-associated drug efflux pump and is thought to be a potential cause of taxane resistance in tumors. Also unlike traditional taxanes, Cabazitaxel has exhibited penetration through the blood-brain barrier (BBB.) Preclinical studies have demonstrated that Cabazitaxel was cytotoxic for cell lines with acquired resistance to doxorubicin, vincristine, vinblastine, paclitaxel or docetaxel.

Taxanes have demonstrated statistically significant antitumor activity as both monotherapy and as part of combination triplet regimens in gastroesophageal carcinoma.Cabazitaxel has emerged as a novel investigational semi-synthetic taxoid that has established activity in cell lines refractory to traditional taxanes in preclinical studies and now in a phase III study in patients with metastatic prostate cancer. Cabazitaxel, with its low affinity for the P-glycoprotein drug efflux pump, may demonstrate superior response rates to docetaxel. Furthermore, as demonstrated in prostate cancer, cabazitaxel appears to have substantial activity in patients who have previously been treated with docetaxel.

Phase I and II trials have been conducted demonstrating safety and efficacy of Cabazitaxel (XRP6258) in metastatic breast and prostate cancer. Neutropenia was the primary dose-limiting toxicity with the recommended dose established at 20 and 25mg/m2. The latter dose was used in the TROPIC trial, the pivotal phase III trial demonstrating improved overall survival and median progression free survival in patients with hormone resistant prostate cancer refractory to docetaxel who had received Cabazitaxel plus prednisone versus those who received mitaxantrone plus prednisone. Cabazitaxel given at IV doses of 25mg/m2 has demonstrated both safety and anti-tumor efficacy in phase I, II and now phase III trials

The primary goal is to evaluate the activity of Cabazitaxel for the treatment of advanced gastroesophageal cancer that has progressed after at least one line of treatment for metastatic disease. Activity will be defined as a complete or partial response. The investigators will differentiate between a 10% level of activity and a 30% level of activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients are required to have histologically or pathologically confirmed metastatic gastric or esophageal adenocarcinoma.
* Patients must demonstrate relapse or progression after at least one prior line of chemotherapy for metastatic disease.
* Patients must have measurable disease by CT scan or MRI
* Absolute neutrophil count ≥ 1,500/uL, platelet ≥ 100,000/uL and Hgb > 8.0 g/dl.
* Total bilirubin ≤ upper institutional limit of normal (ULN), and AST or ALT ≤ 3x ULN; if liver metastases then AST or ALT < 5x ULN
* Peripheral neuropathy must be ≤ Grade 1
* Creatinine < 2 x ULN
* ECOG performance status 0 to 2
* Minimum life expectancy of 12 weeks.
* Age older than 18 years.
* Voluntary, signed written informed consent.
* Women of childbearing potential must have a negative pregnancy test Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.

Exclusion Criteria:

* History of severe hypersensitivity reaction to Cabazitaxel or other drugs formulated with polysorbate 80.
* Patients with known, untreated brain metastasis
* Any uncontrolled severe, intercurrent illness.
* Women who are breast-feeding.
* Patients who have undergone major surgery, chemotherapy, or radiotherapy within the last 3 weeks.
* Patients on concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard safran, MD, Principal Investigator — Brown University
Locations (3):
- United States (3):
  - Memorial Hospital, Pawtucket, Rhode Island
  - Brown University Oncology Research Group, Providence, Rhode Island
  - Roger Williams, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Real Drug
Started | 15 (15 patients were enrolled to the study but only 13 went on to begin treatment)
Completed | 13
Not Completed | 2
Not completed — Progression/worsening of Dx prior to txt | 2

BASELINE CHARACTERISTICS:
Population: Patients with metastatic gastroesophageal cancer that have relapsed after at least one line of chemotherapy
Arm/Group | Real Drug
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (7.9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Without Progression at 3 Months
Description: Response will be assessed via RECIST 1.1 criteria
Time Frame: every three cycles approx every 63 days
Measure: Number; unit: participants
Arm/Group | Real Drug
Number analyzed (Participants) | 13
participants | 11

2. Secondary Outcome: Number of Patients Experienced a Toxicity Associated With Cabazitaxel for Patients With Metastatic Gastroesophageal Adenocarcinomas That Have Progressed After at Least One Line of Therapy for Metastatic Disease.
Description: CTCAE version 4. It is noted that the time frame was approximately 7 months, taking into account the total amount of treatment patients received on this trial.
Time Frame: During treatment and through 30 days post treatment, approximately 7 months
Population: Number of patients who experienced a toxicity on the trial. Not all toxicities may be related to study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Real Drug
Number analyzed (Participants) | 13
Participants | 13

ADVERSE EVENTS:
Arm/Group | Real Drug
Serious Adverse Events (participants affected / at risk) | 5/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real Drug (N=13)
Diarrhea, nausea, vomiting (Investigations) | 1 (1)
neutropenia, fever , weakness (Investigations) | 1 (1) — neutropenia (4), fever (1), weakness(3)
pneumonia and anemia (Investigations) | 1 (1) — pneumonia (4) anemia (3)
pleural effusion (Investigations) | 1 (1) — PE (3)
neutopenia, WBC, febrile neutropenia and fever (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real Drug (N=13)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) — 1 patient experienced grade 1 ANC, 2 patients experienced grade 3 ANC, 2 pts experienced grade 4 ANC
abd pain (Investigations) | 4 (4)
Alk (Investigations) | 1 (1)
Anemia (Investigations) | 12 (12)
barret esophagus (Investigations) | 1 (1)
bone pain (Investigations) | 1 (1)
Ca (Investigations) | 2 (2)
cellulitis (Investigations) | 1 (1)
creatinine (Investigations) | 1 (1)
Diarrhea (Investigations) | 5 (5)
diverticulitis (Investigations) | 1 (1)
dizziness (Investigations) | 1 (1)
dry mouth (Investigations) | 1 (1)
edema (Investigations) | 1 (1)
erythema (Investigations) | 1 (1)
fatigue (Investigations) | 5 (5)
glucose (Investigations) | 6 (6)
Headache (Investigations) | 1 (1)
heartburn (Investigations) | 1 (1)
hypoalbumin (Investigations) | 7 (7)
hypokalemia (Investigations) | 2 (2)
LFTs (Investigations) | 2 (2)
lymphopenia (Investigations) | 2 (2)
Hyponatremia (Investigations) | 1 (1)
nausea (Investigations) | 6 (6)
pain (Investigations) | 1 (1)
proteinuria (Investigations) | 1 (1)
RBC (Investigations) | 3 (3)
rhinitis (Investigations) | 1 (1)
SOB (Investigations) | 1 (1)
cough (Investigations) | 1 (1)
Thrombocytopenia (Investigations) | 5 (5)
Thursh (Investigations) | 1 (1)
Typhilitis (Investigations) | 1 (1)
vomiting (Investigations) | 3 (3)
WBC (Investigations) | 3 (3)
weakness (Investigations) | 1 (1)
wt loss/anorexia (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No